CLINICAL TRIAL: NCT01133574
Title: A Double-Blind, Randomized, Placebo Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles of SLV354 After Oral Dose Administration in Healthy Adult Male Subjects
Brief Title: This is a Single Ascending Dose Tolerance Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part A completed successfully 22 July 2010, Part B will be separate PET study
Sponsor: Abbott (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S354.1.001; 2009-017008-10 (EudraCT Number)
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Cognition Disorders
Keywords: Healthy volunteers; SLV354; Phase I; SRDT
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (14):
- A1 (Experimental): Part A, Parallel design Arm 1
  Interventions: Drug: SLV354 capsules
- A2 (Experimental): Part A, Parallel design Arm 2
  Interventions: Drug: SLV354 capsules
- A3 (Experimental): Part A, Parallel design Arm 3
  Interventions: Drug: SLV354 capsules
- A4 (Experimental): Part A, Parallel design Arm 4
  Interventions: Drug: SLV354 capsules
- A5 (Experimental): Part A, Parallel design Arm 5
  Interventions: Drug: SLV354 capsules
- A6 (Experimental): Part A, Parallel design Arm 6
  Interventions: Drug: SLV354 capsules
- A7 (Experimental): Part A, Parallel design Arm 7
  Interventions: Drug: SLV354 capsules
- A8 (Experimental): Part A, Parallel design Arm 8
  Interventions: Drug: SLV354 capsules
- A9 (Placebo Comparator): Part A, Parallel design Arm 9
  Interventions: Drug: Placebo capsules
- B1-1 (Experimental): Part B, Cross-over design, Arm 1
  Interventions: Drug: SLV354 capsules
- B1-2 (Experimental): Part B, Cross-over design, Arm 2
  Interventions: Drug: SLV354 capsules
- B2-1 (Experimental): Part B, Cross-over design, Arm 3
  Interventions: Drug: SLV354 capsules
- B2-2 (Experimental): Part B, Cross-over design, Arm 4
  Interventions: Drug: SLV354 capsules
- B3 (Placebo Comparator): Part B, Cross-over design, Arm 5
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: SLV354 capsules — 20 mg
  Arms: A1
Drug: SLV354 capsules — 60 mg
  Arms: A2
Drug: SLV354 capsules — 120 mg
  Arms: A3
Drug: SLV354 capsules — 250 mg
  Arms: A4
Drug: SLV354 capsules — 500 mg
  Arms: A5
Drug: SLV354 capsules — 750 mg
  Arms: A6
Drug: SLV354 capsules — 1000 mg
  Arms: A7
Drug: SLV354 capsules — 1250 mg
  Arms: A8
Drug: Placebo capsules — placebo
  Arms: A9
Drug: SLV354 capsules — low dose group 1
  Arms: B1-1
Drug: SLV354 capsules — high dose group 1
  Arms: B1-2
Drug: SLV354 capsules — low dose group 2
  Arms: B2-1
Drug: SLV354 capsules — high dose group 2
  Arms: B2-2
Drug: Placebo capsules — placebo
  Arms: B3

SUMMARY:
This is a single rising dose tolerance (Part A) followed by a functional magnetic resonance imaging (Part B)

DETAILED DESCRIPTION:
The Part A of this study is a parallel design followed in a second part by a cross-over design

ELIGIBILITY:
Inclusion Criteria

* BMI 18.0 to 28.0 kg/m2,
* systolic blood pressure 90-140 mmHg,
* diastolic blood pressure 50-90 mmHg,
* heart rate 50 100 beats/min (all inclusive),
* clinically normal safety ECG and laboratory results

Exclusion Criteria

* relevant disease,
* treated with SLV354 before

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments including adverse events, clinical laboratory tests, ECG and vital signs (Part A) | 1 week after each dose level
Safety and tolerability assessments including adverse events, clinical laboratory tests, ECG and vital signs (Part B) | 2 weeks after each dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters (AUC and Cmax) after single ascending oral dosing of max. 8 doses of SLV354 ranging from 20 to 1250 mg (Part A) | 1 week after each dose level
Pharmacodynamic variables (EEG, Cognitive tests, Questionnaires, plasma hormones ACTH / cortisol / TSH / T3 / T4) (Part A) | 1 week after each dose level
Pharmacokinetic parameters (AUC and Cmax) after single oral dosing of 2-4 doses of SLV354 chosen (Part B) | 2 weeks after each dose
Pharmacodynamic variables : Cognitive tests, Questionnaires, fMRI) (Part B) | 2 weeks after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Rendenbach-Mueller, PhD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 62002, London, United Kingdom